CLINICAL TRIAL: NCT01821677
Title: A Randomized, Placebo-Controlled, Parallel, Double-Masked Study to Evaluate the Efficacy and Safety of Two Doses of Oral Optina™ in Adult Patients With Diabetic Macular Edema
Brief Title: A Safety and Efficacy Study of Oral Danazol (a Previously Approved Drug) in the Treatment of Diabetic Macular Edema.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ampio Pharmaceuticals. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AP-05-002
Record Dates: First submitted 2013-03-25; First posted 2013-04-01 (Estimated); Results first posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-08

CONDITIONS: Diabetic Macular Edema
Keywords: macular edema; diabetic
MeSH Terms: conditions — Macular Edema | interventions — Danazol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low Dose Danazol (Experimental): Capsules, 0.5 mg/BMI Danazol with dose determined by subject's BMI at baseline, 2 capsules (5 mg, 7.5 mg, or 10 mg) twice daily, for 12 weeks.
  Interventions: Drug: Danazol Capsules
- High Dose Danazol (Experimental): Capsules, 1.0 mg/BMI Danazol with dose determined by subject's BMI at baseline, 2 capsules (5 mg, 7.5 mg, or 10 mg) twice daily, for 12 weeks.
  Interventions: Drug: Danazol Capsules
- Placebo (Placebo Comparator): Gelatin capsules, identical in appearance to the active capsules, filled with pharmaceutical grade lactose and magnesium stearate.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Danazol Capsules
  Other Names: Optina; Cyclomen; Danocrine
  Arms: High Dose Danazol; Low Dose Danazol
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy of ultra low dose danazol (Optina™) for the treatment of diabetic macular edema.

DETAILED DESCRIPTION:
A Randomized, Placebo-Controlled, Parallel, Double-Masked Study to Evaluate the Efficacy and Safety of Two Doses of Oral Optina™ in Adult Patients With Diabetic Macular Edema.

The primary trial objective is to evaluate the efficacy of two oral BMI-related doses (0.5 mg per body mass index (BMI), 1.0 mg per BMI per day) of Optina™ in improving visual acuity (VA) compared to placebo.

The secondary objectives are to evaluate the efficacy of two oral BMI-related doses of Optina™ on change in central macular thickness (CMT) and VA responder status compared to placebo, and to assess the safety and tolerability of two oral BMI-related doses of Optina™ compared to placebo.

ELIGIBILITY:
Study Level Inclusion Criteria:

1. Subject is willing and able to provide informed consent for study participation
2. Male or female 18 years or older with Type 1 or 2 diabetes mellitus [defined as a self-report of diabetes accompanied by treatment (insulin or diet) or a history of fasting plasma glucose ≥ 7.0 mmo/l (126 mg/dl) or 2-hr plasma glucose ≥ 11.1 mmo/l (200 mg/dl)]
3. Female subjects of childbearing potential must have a negative pregnancy test within 7 days prior to randomization and must agree to utilize a reliable form of effective contraception (hormonal or barrier method; abstinence) throughout the study and for 90 days after the last dose of study medication. Childbearing potential is defined as women who have had menses within the past 12 months, who have not had tubal ligation or bilateral oophorectomy [Note: patients using contraceptive methods containing progesterone (including a progesterone IUD) for 90 days prior to randomization or planning to use progesterone contraceptive methods (including a progesterone IUD) during the study drug treatment period are not eligible for enrollment.] Should a woman become pregnant or suspect that she is pregnant while participating in this study, she should inform her treating physician immediately
4. Enrollment in this study is contraindicated for pregnant or lactating women. Thus, female patients who are postmenopausal without a menstrual period for ≥ 12 months, surgical sterility, not pregnant and not breast feeding for 90 days prior to randomization can be enrolled
5. At least one eye meets the study eye criteria for inclusion in the study (see Study Eye Inclusion Criteria, below)
6. Stable diabetic and metabolic control (no major changes in diabetic or lipid reducing medications for 3 months prior to start of this study as determined by the Investigator)

Study Eye Inclusion Criteria (if both eyes meet criteria, both eyes will be study eyes)

1. Change in VA within previous 12 months reasonably believed to be associated with diabetic macular edema (DME) in the opinion of the Investigator
2. Best-corrected visual acuity (BCVA) in accordance with early treatment diabetic retinopathy study (ETDRS) letter score of ≥24 (e.g., 20/320 or better) and ≤78 (e.g., 20/32 or worse)
3. Definite retinal thickening ≥275 microns on spectral-domain optical coherence tomography (OCT) due to DME involving the center of the macula on clinical exam in the opinion of the Investigator
4. Media clarity, pupillary dilation, and patient cooperation sufficient for adequate fundus photographs
5. Assessment by the Investigator that focal photocoagulation can be deferred safely for 16 weeks

Study Level Exclusion Criteria:

1. Known allergy to any danazol (Cyclomen® or Danocrine®) or any other non-medicinal component of the danazol test drug (cornstarch, lactose, magnesium stearate, gelatin, and talc) (Note: Lactose intolerance is not a contraindication to ingesting the small amount of lactose contained in oral medications)
2. Known allergy to any component of the placebo test drug (lactose, magnesium stearate, and gelatin)
3. History of systemic (e.g., oral, intravenous, intramuscular, subcutaneous, intra-uterine, epidural, bursal, or implanted) androgens, progesterone or corticosteroids (including topical ophthalmic corticosteroids preparations within 4 months prior to randomization (topical non-ophthalmic corticosteroids are not excluded)
4. Blood pressure >180/110 mm Hg (in cases where either or both of the systolic or diastolic limits are exceeded, blood pressure can be re-measured after 10 minutes rest period for inclusion in the study)
5. HbA1c greater than 11% or consistent HbA1c values in a similar range for the last 6 months.
6. Carcinoma of the breast
7. Prostate cancer
8. Androgen-dependent tumor
9. Undiagnosed abnormal genital bleeding
10. Genital neoplasia
11. Currently taking warfarin (coumadin), carbamazepine, phenytoin, phenobarbital cyclosporin or tacrolimus
12. Females who are pregnant or planning pregnancy in the 6-month period after randomization (Note: Enrollment in this study is contraindicated for pregnant or lactating women)
13. Females breast feeding or breast feeding in the 90 days prior to randomization (Note: Enrollment in this study is contraindicated for pregnant or lactating women)
14. Use of any hormonal therapies including hormone replacement therapy (HRT) and contraceptive medications that contain progesterone within 3 months before randomization (Note: patients on pure estrogen or estradiol replacement therapy can be enrolled in the study)
15. Unstable cardiovascular disease or a history of significant heart disease (including unstable angina, acute coronary syndrome, myocardial infarction, or history of coronary revascularization procedure) within 6 months before randomization
16. Any condition that, in the opinion of the Investigator, would preclude participation in the study (e.g., unstable medical status including blood pressure and glycemic control). Patients in poor glycemic control who, within the last 3 months, using a new type of insulin (for example, changing to or adding a short acting insulin from a longer-acting insulin), or increased the daily dose ≥ 50%, initiated intensive insulin treatment such as an insulin pump or additional daily injections or plan to do so in the next 3 months should not be enrolled.
17. Significant hepatic disease (defined as aspartate aminotransferase, alanine aminotransferase or alkaline phosphatase [ALP], more than twice the upper limit of normal) where, in the opinion of the Investigator, danazol might be contraindicated
18. Significant renal disease (defined as serum creatinine ≥ 2.5 mg/dl, history of renal transplant, or undergoing dialysis at screening) where, in the opinion of the Investigator, danazol might be contraindicated
19. Changes in anti-hypertensive medication within 3 months before randomization (except for dosage adjustments that are considered minor in the opinion of the Investigator)
20. Major surgery (e.g., head and neck, chest, abdomen, gastrointestinal, genitourinary or central nervous system) within past 28 days or anticipated in the next 6 months
21. History of acute intermittent porphyria, any thrombosis or thromboembolic disease or pseudotumor cerebri
22. Participation in an investigational trial within 30 days of study entry that involved treatment with any drug that has not received regulatory approval at the time of study entry
23. Patient is expecting to move out of the area of the clinical center during the next 6 months

Study Eye Exclusion Criteria:

1. Macular edema considered to be due to a cause other than DME; e.g., cataract extraction, vitreo-retinal interface disease (a taut posterior hyaloid or epiretinal membrane)
2. An ocular condition is present such that, in the opinion of the Investigator, VA would not improve from resolution of macular edema (e.g., foveal atrophy, closure of juxtafoveal capillaries, dense subfoveal hard exudates)
3. An ocular condition (other than diabetic retinopathy) that, in the opinion of the Investigator, might affect macular edema or alter VA during the course of the study, e.g., vein occlusion, uveitis or other ocular inflammatory disease, Irvine-Gass Syndrome, etc.
4. Substantial cataract that, in the opinion of the Investigator, is likely to interfere with ocular measurements or evaluations during this study
5. History of treatment for DME at any time in the past 8 weeks (such as focal/grid macular photocoagulation, intravitreal or peribulbar corticosteroids, anti-vascular endothelial growth factor [VEGF drugs], or any other treatment). Note, the 28-day screening period allows subjects to be screened at 4 weeks post DME treatment and have a baseline visit 28 days later.
6. History of panretinal scatter photocoagulation (PRP) within 4 months prior to randomization or anticipated need for PRP in the 6 months following randomization
7. History of major ocular surgery (including cataract extraction, scleral buckle, any intraocular surgery, etc.) within prior 6 months or anticipated within the next 6 months following randomization
8. History of yttrium aluminum garnet (YAG) capsulotomy performed within 2 months prior to randomization
9. Uncontrolled glaucoma (in Investigator's judgment) in the study eye
10. Aphakia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2013-02-26 (Actual); Primary Completion 2014-10-30 (Actual); Study Completion 2015-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Levy, M.D., Study Director — Ampio Pharmaceuticals. Inc.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bar-Or D, Orlando A, Singer M; danazol study group. Potential beneficial effect of low-dose danazol in combination with renin-angiotensin system inhibitors in diabetic macular oedema. Acta Ophthalmol. 2017 Nov;95(7):e665-e667. doi: 10.1111/aos.13318. Epub 2016 Nov 19. No abstract available. PMID 27864867

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited for study enrollment from a population of subjects being seen by clinicians participating in the investigational trial. Recruitment occurred from February 2013 to June 2014.
Pre-assignment Details: Standard of care treatment for diabetes will not be withheld during the study.
Units Other Than Participants: Eyes
Groups:
- Low Dose Danazol: Low Dose Danazol 0.5 mg / BMI administered as 2 capsules twice daily (total of 4 capsules/day) for 12 weeks.
- High Dose Danazol: High Dose Danazol 1.0 mg / BMI administered as 2 capsules twice daily (total of 4 capsules/day) for 12 weeks.
- Placebo: Placebo (lactose and magnesium stearate) administered as 2 capsules twice daily (total of 4 capsules/day) for 12 weeks.
Period: Overall Study
Arm/Group | Low Dose Danazol | High Dose Danazol | Placebo
Started | 117; 141 Eyes | 117; 142 Eyes | 120; 142 Eyes
Completed | 94; 114 Eyes | 102; 126 Eyes | 105; 124 Eyes
Not Completed | 23; 27 Eyes | 15; 16 Eyes | 15; 18 Eyes
Not completed — Adverse Event | 4 | 6 | 5
Not completed — Physician Decision | 1 | 4 | 1
Not completed — Non-compliance | 0 | 1 | 2
Not completed — Lost to Follow-up | 2 | 1 | 3
Not completed — Protocol Violation | 0 | 0 | 2
Not completed — Withdrawal by Subject | 7 | 3 | 2
Not completed — Other | 9 | 0 | 0

BASELINE CHARACTERISTICS:
Population: If both eyes met the study eye inclusion criteria, both eyes were used as study eyes.
Units Other Than Participants: Eyes
Groups:
- Low Dose Danazol: 0.5 mg/BMI/day of Danazol administered as 2 capsules twice daily (total of 4 capsules/day) for 12 weeks.
- High Dose Danazol: 1.0 mg/BMI/day of Danazol administered as 2 capsules twice daily (total of 4 capsules/day) for 12 weeks.
- Placebo: Placebo capsules administered as 2 capsules twice daily (total of 4 capsules/day) for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Low Dose Danazol | High Dose Danazol | Placebo | Total
Number analyzed (Participants) | 117 | 117 | 120 | 354
Number analyzed (Eyes) | 141 | 142 | 142 | 425
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.2 (11.2) | 62.7 (8.8) | 62.4 (10.6) | 63.1 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 51 | 68 | 177
  Male | 59 | 66 | 52 | 177
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 27 | 31 | 86
  Not Hispanic or Latino | 89 | 90 | 89 | 268
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 0 | 3
  Asian | 2 | 2 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 3 | 1 | 0 | 4
  Black or African American | 13 | 10 | 7 | 30
  White | 97 | 102 | 109 | 308
  More than one race | 1 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 117 | 117 | 120 | 354
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 32.3 (7.1) | 32.2 (6.9) | 32.3 (6.8) | 32.3 (6.9)
Best Corrected Visual Acuity (BCVA) [Mean (Standard Deviation); unit: Letters Correctly Read] — Letters read in accordance with Early Treatment Diabetic Retinopathy Study (ETDRS) at Baseline
  Letters Correctly Read | 63.8 (11.2) | 63.6 (10.2) | 62.7 (11.6) | 63.4 (11.0)
Central Macular Thickness [Mean (Standard Deviation); unit: micrometers (μm)] — Center subfield retinal thickness as measured by optical coherence tomography (OCT) at Baseline Population: Number of eyes analyzed differs from overall population
  micrometers (μm) | 438.6 (132.8) | 423.3 (120.8) | 426.8 (126.9) | 430.1 (127.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Best Corrected Visual Acuity (BCVA)
Description: Change from baseline score to the week 12 score in the number of letters read on an eye chart in accordance with Early Treatment Diabetic Retinopathy Study (ETDRS) of the Intent to Treat (ITT) population of all treated subjects. A positive number indicates more letters could be read.
Time Frame: Determined at Baseline and Week 12
Population: Intent to Treat (ITT)
Measure: Mean (95% Confidence Interval); unit: Letters Correctly Read
Units Other Than Participants: Eyes
Groups:
- Danazol Combined (0.5 mg / BMI and 1.0 mg / BMI Dose): Combined Results of 0.5 mg / BMI (Low) and 1.0 mg / BMI (High) Dose administered as 2 capsules twice daily (total of 4 capsules/day) for 12 weeks.
Arm/Group | Low Dose Danazol | High Dose Danazol | Danazol Combined (0.5 mg / BMI and 1.0 mg / BMI Dose) | Placebo
Number analyzed (Participants) | 117 | 117 | 234 | 120
Number analyzed (Eyes) | 141 | 142 | 283 | 142
Letters Correctly Read | 1.0 [-0.3 to 2.4] | 0.8 [-0.4 to 2.0] | 0.9 [0.0 to 1.8] | 2.5 [1.5 to 3.5]
Statistical Analysis 1: Comparison: Low Dose Danazol vs Placebo; Test type: Superiority; p = 0.16, ANCOVA
Statistical Analysis 2: Comparison: High Dose Danazol vs Placebo; Test type: Superiority; p = 0.07, ANCOVA
Statistical Analysis 3: Comparison: Danazol Combined (0.5 mg / BMI and 1.0 mg / BMI Dose) vs Placebo; Test type: Superiority; p = 0.03, ANCOVA

2. Secondary Outcome: Change in Central Macular Thickness (CMT)
Description: A measured change from baseline to week 12 of central macular thickness of the Intent to Treat population of all treated subjects. A negative difference in Central Macular Thickness constitutes a reduction in retinal thickness. Increase in Central Macular Thickness is caused by diabetic macular edema. A greater negative value indicates a greater reduction in swelling.
Time Frame: Determined at Baseline and Week 12
Population: Intent to Treat (ITT)
Measure: Mean (95% Confidence Interval); unit: micrometers (μm)
Units Other Than Participants: Eyes
Arm/Group | Low Dose Danazol | High Dose Danazol | Danazol Combined (0.5 mg / BMI and 1.0 mg / BMI Dose) | Placebo
Number analyzed (Participants) | 117 | 117 | 234 | 120
Number analyzed (Eyes) | 141 | 142 | 283 | 142
micrometers (μm) | -6.0 [-20.5 to 8.6] | -2.8 [-17.6 to 12.00] | -4.4 [-14.7 to 5.9] | -17.5 [-33.1 to -2.0]
Statistical Analysis 1: Comparison: Low Dose Danazol vs Placebo; Test type: Superiority; p = 0.42, ANCOVA
Statistical Analysis 2: Comparison: High Dose Danazol vs Placebo; Test type: Superiority; p = 0.28, ANCOVA
Statistical Analysis 3: Comparison: Danazol Combined (0.5 mg / BMI and 1.0 mg / BMI Dose) vs Placebo; Test type: Superiority; p = 0.14, ANCOVA

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: Patients will be followed for all adverse events (AEs) until 30 days after the last dose of study medication. All AEs considered to be possibly related to Optina™ will be followed until the event resolves or stabilized without further change. Adverse events were assessed by participant level not eyes (units analyzed).
Groups:
- Low Dose Danazol: Low Dose Danazol 0.5 mg / BMI
- High Dose Danazol: High Dose Danazol 1.0 mg / BMI
- Placebo: Placebo (lactose and magnesium stearate)
Arm/Group | Low Dose Danazol | High Dose Danazol | Placebo
All-Cause Mortality (participants affected / at risk) | 1/117 | 0/117 | 0/120
Serious Adverse Events (participants affected / at risk) | 14/117 | 7/117 | 12/120
Other Adverse Events (participants affected / at risk) | 32/117 | 34/117 | 48/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose Danazol (N=117) | High Dose Danazol (N=117) | Placebo (N=120)
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0 | 0
Angina Unstable (Cardiac disorders) | 1 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 1
Cardiac Arrest (Cardiac disorders) | 1 | 0 | 0
Cardiac Failure Chronic (Cardiac disorders) | 1 | 0 | 0
Cardiac Failure Congestive (Cardiac disorders) | 1 | 1 | 0
Coronary Artery Occlusion (Cardiac disorders) | 0 | 1 | 1
Diabetic Retinopathy (Eye disorders) | 0 | 0 | 1
Glaucoma (Eye disorders) | 0 | 1 | 1
Vitreous Haemorrhage (Eye disorders) | 0 | 0 | 1
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Oedema Peripheral (General disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0
Gas Gangrene (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Localised Infection (Infections and infestations) | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Metabolic Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Colorectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 0 | 0
Diabetic Como (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Nephropathy (Renal and urinary disorders) | 1 | 0 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 1 | 1
Ureteric Stenosis (Renal and urinary disorders) | 0 | 0 | 1
Ovarian Mass (Reproductive system and breast disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose Danazol (N=117) | High Dose Danazol (N=117) | Placebo (N=120)
Vitreous Haemorrhage (Eye disorders) | 7 | 5 | 8
Diabetic Retinal Oedema (Eye disorders) | 2 | 7 | 5
Hypertension (Vascular disorders) | 5 | 4 | 5
Nausea (Gastrointestinal disorders) | 3 | 2 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 5
Eye Pain (Eye disorders) | 2 | 2 | 3
Headache (Nervous system disorders) | 2 | 4 | 1
Nasopharyngitis (Infections and infestations) | 3 | 2 | 2
Oedema Peripheral (General disorders) | 3 | 1 | 3
Urinary Tract Infection (Infections and infestations) | 1 | 1 | 5
Sinusitis (Infections and infestations) | 4 | 1 | 1
Vitreous Detachment (Eye disorders) | 0 | 2 | 3
Dry Eye (Eye disorders) | 0 | 1 | 3

LIMITATIONS AND CAVEATS:
The study may have been underpowered to detect a difference in certain endpoints in some arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes